CLINICAL TRIAL: NCT06145269
Title: Recanalization Rate of Acute Deep Venous Thrombosis Related to Therapeutic Modality- Comparative Study; New Oral Anticoagulants (NOACs) Vs. Conventional Treatment.
Brief Title: Recanalization Rate of Acute DVT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mahmoud Yaseen, Assistant Lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Recanalization rate(acute DVT)
Record Dates: First submitted 2023-11-13; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Acute DVT of Lower Extremity
MeSH Terms: interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New oral anticoagulant (rivaroxaban) (Active Comparator): We will use (rivaroxaban) 15 mg oral tablets twice a day, After 21 days: Should transition to 20 mg orally once a day untill we complete 6 months from the starting the treatment.
  Interventions: Drug: New oral anticoagulant (rivaroxaban) and Marevan (warfarin)
- Marevan (warfarin) (Active Comparator): Initiate warfarin on day 1 or 2 of parenteral anticoagulation therapy (eg, LMWH or unfractionated heparin) Overlap warfarin and parenteral anticoagulant for at least 5 days until desired INR (>2.0) maintained for 24 hours, then discontinue parenteral therapy and continue only with (warfarin) tablets 5 mg/day for 6 months.
  Interventions: Drug: New oral anticoagulant (rivaroxaban) and Marevan (warfarin)

INTERVENTIONS:
Drug: New oral anticoagulant (rivaroxaban) and Marevan (warfarin) — comparison between 2 drug, (rivaroxaban) and Marevan (warfarin)

SUMMARY:
Rporting and evaluation of the rate of recanalization of acute DVT of the lower limb at one year follow-up comparing the results of using NOACs vs. conventional treatment.

DETAILED DESCRIPTION:
Deep vein thrombosis (DVT) is an important cause of disability and mortality in our society . The incidence of DVT significantly increases with age, being more prevalent in women than men . The location of DVT is also an important factor to be studied because of its association with pulmonary embolism and development of post-thrombotic syndrome (PTS) , Currently, duplex ultrasound scanning (DUS) is the method of choice for diagnosis of DVT because it is non-invasive, provides real-time imaging, and has high sensitivity and specificity especially for detection of proximal DVT .

The new oral anticoagulants (NOACs), are poised to replace warfarin for treatment of the majority of patients with venous thromboembolism (VTE), With a rapid onset of action and the capacity to be administered in fixed doses without routine coagulation monitoring, NOACs have been shown to be noninferior to conventional anticoagulant therapy for prevention of recurrence with less bleeding.

Most studies have reported that more advantages than disadvantages for NOACs when compared with VKAs, with the most important advantages of NOACs including safety issues (ie, a lower incidence of major bleeding), convenience of use, minor drug and food interactions, a wide therapeutic window, and no need for laboratory monitoring. Nonetheless, there are some conditions for which VKAs remain the drug of choice.

ELIGIBILITY:
Inclusion Criteria:

* • Patients suffering from first attack of acute DVT (De novo) of the lower limb who (only femoral-popliteal type) aged 18 - 80 years.

Exclusion Criteria:

* Patients suffering from recurrent DVT.
* Patients with acute DVT candidate for CDT (limb threatening acute DVT).
* Patients suffering from acute DVT with malignancy.
* Pregnant and Lactating females.
* Patients with severe renal Impairment (CrCl <30mL/min), Severe hepatic impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Recanalization rate of the thrombosed vein with the two comparable groups. | baseline
  Reporting and evaluation the rate of recanalization of acute DVT of the lower limb at one year follow-up comparing the results of using NOACs vs. conventional treatment.

REFERENCES:
- See also: INCIDENCE OF DEEP VENOUS THROMBOSIS IN STROKE PATIENTS IN MEDICAL INTENSIVE CARE UNIT ZAGAZIG UNIVERSITY HOSPITALS, EGYPT — http://zumj.journals.ekb.eg/article_4349_5855d1034c50f928ccadc9384e6d656c.pdf